CLINICAL TRIAL: NCT03589547
Title: Durvalumab and Consolidation SBRT Following Chemoradiation for Locally Advanced Stage III Non-Small Cell Lung
Acronym: 358
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Lifespan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG 358
Record Dates: First submitted 2018-06-22; First posted 2018-07-18 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Stage III Non-small-cell Lung Cancer
Keywords: Lung cancer; NSCLC; Stage III; Post chemoradiation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — durvalumab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Durvalumab and SBRT (Experimental): Durvalumab 10mg/kg x 1 day, dose #1 to occur > 3 weeks and <7 weeks after last chemo/RT and prior to SBRT dose 1 (5-10 day time frame between Durvalumab and SBRT).
  SBRT boost will consist of 2 fractions delivered to the primary tumor only, over 1-2 weeks between the first and second treatments with durvalumab (see above for time frames). The dose will consist of 20Gy (2 fractions of 10Gy). 3 fractions are allowed for centrally located tumors
  Dose # 2 of durvalumab, (post SBRT) to be given 1-10 days post last SBRT. Durvalumab then to be given at 10mg/kg Q2 weeks (+/- 4 days) for a total of 12 months (maximum of 26 treatments total)
  Interventions: Drug: Durvalumab; Radiation: SBRT

INTERVENTIONS:
Drug: Durvalumab — Durvalumab10mg/kg Q2 weeks (+/- 4 days) for a total of 12 months (maximum of 26 treatments total)
  Other Names: Imfinzi
Radiation: SBRT — SBRT boost will consist of 2 fractions delivered to the primary tumor only, over 1-2 weeks between the first and second treatments with durvalumab.
  The dose will consist of 20Gy (2 fractions of 10Gy)
  *3 fractions are allowed for centrally located tumors
  Other Names: Stereotactic body radiation

SUMMARY:
Durvalumab is a drug that stimulates the immune system to fight lung cancer. Durvalumab is FDA approved to treat lung cancer. Stereotactic body radiation therapy (SBRT) is a newer radiation treatment that gives fewer, but higher doses of radiation than standard radiation.

With SBRT, radiation is focused toward the cancer and away from normal surrounding lung tissue. It is possible that when cancer cells are damaged by SBRT Durvalumab may be more effective in activating the immune system. SBRT is a standard FDA approved treatment for early stage (stage 1) lung cancer and is investigational in patients such as yourself with stage 3 lung cancer. The combination of Durvalumab and SBRT is investigational. This study will investigate the effects, good and bad, of the combination of Durvalumab and SBRT.

ELIGIBILITY:
Inclusion Criteria:

* Stage III NSCLC.
* Completion of concurrent chemoradiation:

  • Radiation dose of 60.0 Gy (50-65Gy) using standard fractionation
* Patients will receive the first dose of durvalumab > 3 weeks and < 7 weeks after their last treatment of chemoradiation (last radiation or chemotherapy treatment, whichever ended last).Sites are required to submit prior treatment (chemotherapy and radiation)
* Residual tumor volume that is appropriate for SBRT

  • Residual Primary tumor <120cc (approximately 6cm diameter).
* Absolute neutrophil count ≥ 1,000/uL, platelet ≥ 60,000/uL prior to registration.
* Total bilirubin ≤ 1.5x upper institutional limit of normal (ULN), and AST and ALT ≤ 3x ULN.
* ECOG performance status 0 to 1
* Minimum life expectancy of 12 weeks as determined by treating physician.
* Age > 18 years.
* Voluntary, signed written informed consent.
* Women of childbearing potential must have a negative serum pregnancy test within 7 days of day 1 of treatment (post-menopausal women, defined as surgical menopause or lack or menses >12 months, do not need to have a pregnancy test, document status.)
* Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 6 months after the last treatment.
* Resolution of all related toxicities from chemo/RT to < grade 2, except alopecia.
* Patient must have tissue available from prior biopsy for correlative studies as confirmed by treating physician.

Exclusion Criteria:

* Disease progression during or after standard chemoradiation
* Prior thoracic radiation (other than the chemoradiation delivered prior to SBRT)
* Metastatic disease
* Uncontrolled severe, intercurrent illness as confirmed by the treating physician.
* Chemotherapy within 3 weeks from the first treatment on study (day 1).
* Prior complete resection of all NSCLC (patients could have undergone prior resection as long as it is not complete and the patient meets criteria and staging and tumor volume for registration).
* Severe, active co-morbidity, defined as follows:

  * Uncontrolled neuropathy ≥ grade 2 regardless of cause;
  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months;
  * Transmural myocardial infarction within the last 6 months;
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration;
  * Severe hepatic disease, defined as a diagnosis of Child-Pugh Class B or C hepatic disease.
  * HIV positive with CD4 count < 200 cells/microliter. Note that patients who are HIV positive are eligible, provided they are under treatment with highly active antiretroviral therapy (HAART) and have a CD4 count ≥ 200 cells/microliter within 30 days prior to registration. Note also that HIV testing is not required for eligibility for this protocol unless patient is known to be HIV positive and they do not had a CD4 count result within 30 days prior to registration.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment, not inclusive of patients who are HIV positive and who meet criterion above.

Note: Patients who require continuous or intermittent steroid therapy for non-autoimmune conditions, e.g. asthma, osteoarthritis or intravenous contrast allergy, are eligible permitted those patients who receive continuous steroids are limited to a dose of ≤10 mg/day of prednisone (or equivalent). Higher doses are permitted for intermittent therapy, e.g. for contrast allergy, but will need to be approved by BrUOG prior to registration.

* Has a known history of active tuberculosis
* Hypersensitivity to Durvalumab or any of its excipients
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has known history of clinically significant pneumonitis
* Has an active infection requiring intravenous systemic therapy at the time of registration
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating physician
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial as per the treating physician
* Is pregnant or breastfeeding
* Has received prior therapy with an anti-CTLA-4, -PD-1, -PD-L1, or -PD-L2 agent
* Has a known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients experiencing grade 2 or higher toxicities during consolidation SBRT with concurrent durvalumab after chemoradiation for locally advanced stage III NSCLC | Defined as the first 3 months of durvalumab.
  This outcome will examine the safety and tolerability of the trial.
Average progression-free survival of chemoradiation followed by SBRT and durvalumab for patients with locally advanced stage III NSCLC. | Every 3 months for 1 year then every 4 months for two years then every 6 months for two years then annually until progression on average for about 5 years.
  RECIST 1.1

SECONDARY OUTCOMES:
Overall survival (OS) | Every 2 months for the first 6 months, then every 4 months for 2 years then every 6 months for 2 years then yearly for about 5 years
Average time to local-regional progression (LRP) | Every 3 months for 1 year then every 4 months for two years then every 6 months for two years then annually until progression for about 5 years.
Time to distant metastasis (DM) | Every 3 months for 1 year then every 4 months for two years then every 6 months for two years then annually until progression.

CONTACTS AND LOCATIONS:
Overall Officials: Hina Khan, MD, Principal Investigator — Brown University Oncology Research Group (BrUOG) & Lifespan Cancer Institute
Locations (2):
- United States (2):
  - Rhode Island Hospital, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island